CLINICAL TRIAL: NCT05792137
Title: Western Human Nutrition Research Center (WHNRC) Postprandial Monocyte Study
Brief Title: Postprandial Monocyte Study
Acronym: PPMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA, Western Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 1999385
Record Dates: First submitted 2023-03-15; First posted 2023-03-31 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Immune System; Nutrition; Inflammation
Keywords: monocyte; postprandial; nonclassical monocytes
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High saturated fat challenge meal followed by high mono-unsaturated fat challenge meal (Experimental): High saturated fat mixed macronutrient challenge meal with palm oil followed by high mono-unsaturated fat mixed macronutrient challenge meal with olive oil two weeks later
  Interventions: Other: High saturated fat challenge meal; Other: High mono unsaturated fat challenge meal
- High mono-unsaturated fat challenge meal followed by high saturated fat challenge meal (Experimental): High mono-unsaturated fat mixed macronutrient challenge meal with olive oil followed by high saturated fat mixed macronutrient challenge meal with palm oil two weeks later
  Interventions: Other: High saturated fat challenge meal; Other: High mono unsaturated fat challenge meal

INTERVENTIONS:
Other: High saturated fat challenge meal — High saturated fat challenge meal made with palm oil
Other: High mono unsaturated fat challenge meal — High mono unsaturated fat challenge meal made with olive oil

SUMMARY:
The purpose of this research is to determine the role of a type of immune cell in blood, called a non-classical monocytes (NCMs), following consumption of a high-fat meal. Previous studies have found that monocytes are important for blood vessel health. In this study, two different high-fat meals will be used to study the effect of different types of dietary fat on postprandial NCMs. The investigators will characterize NCMs in both fasting conditions and following consumption of two different high-fat meals, and will evaluate whether the type of fat in a meal affects NCMs in blood.

DETAILED DESCRIPTION:
Monocytes are a heterogeneous population of circulating blood cells that contribute to tissue integrity as well as to innate and adaptive immune defense. There are three well-characterized subsets based on their relative expression of surface antigens, cluster of differentiation 14 (CD14) and cluster of differentiation 16 (CD16). Monocytes originate from myeloid precursors in the bone marrow and enter the circulation as classical monocytes (CLMs). CLMs represent a transient cell population with a diverse differentiation potential. CLMs comprise 80-90% of the circulating blood monocyte pool and remain in circulation for approximately one day before either migrating into tissue to repopulate the tissue resident macrophage population or maturing into non-classical monocytes (NCMs). NCMs comprise only 5-10% of the circulating blood monocyte pool but have a much longer circulating lifespan of approximately 7 days. NCMs exhibit conflicting functions as anti-inflammatory caretakers of vascular tissue and as contributors to the pathogenesis of disease.

Metabolic responses to food consumption influence the risk of cardiometabolic disease. Postprandial glycemia and lipemia modulate vascular health by altering endothelial function and inducing oxidative stress, inflammation, and apoptosis. Consumption of a single high-fat meal increases circulating interleukin 6 (IL-6), enhances expression of monocyte adhesion molecules, reduces flow-mediated dilation, and increases markers of oxidative stress in human subjects. Although NCMs are described as vascular housekeepers with distinct motility and crawling patterns allowing them to actively surveil endothelium and scavenge luminal debris, their role in the postprandial state is currently unknown.

To better understand the function of postprandial NCMs following consumption of a single high-fat mixed macronutrient challenge meal, the investigators propose a study following a crossover design in which participants will consume one of two isocaloric high-fat challenge meals spaced two-weeks apart, a high-saturated fat mixed macronutrient challenge meal or a high-monounsaturated fat mixed macronutrient challenge meal. Blood at fasting and at six hours postprandial will be collected and the proportion of NCMs and their integrin expression will be analyzed by flow cytometry while changes in global gene expression will be measured by RNA-sequencing.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18.5 - 29.9 kg/m²
* have a bank account and social security number or taxpayer identification for financial compensation

Exclusion Criteria:

* Pregnant or lactating women
* Known allergy or hindering intolerance to study meal ingredients
* Systolic blood pressure greater than 140 mmHg or diastolic blood pressure greater than 90 mmHg measured
* Fasting glucose above 105 mg/dL
* Triglycerides above 150 mg/dL
* HDL cholesterol less than 40 mg/dL (men) and 50 mg/dL (women)
* Self-reported history of difficulties with blood drawing procedures including prior fainting or dizziness, or veins assessed as not suitable for four separate venipunctures by licensed phlebotomist
* Diagnosed active chronic diseases for which the individual is currently taking daily medication, including but not limited to Diabetes mellitus, Cardiovascular disease, Cancer, Gastrointestinal disorders, Kidney disease, Liver disease, Bleeding disorders, Asthma, Autoimmune disorders, Hypertension, Osteoporosis
* Recent minor surgery (within 4 wk) or major surgery (within 16 wk)
* History of gastrointestinal surgery, including gastric bypass surgery or resection
* Recent antibiotic therapy (within 4 wk)
* Known gallbladder disease or history of cholecystectomy
* Recent hospitalization (within 4 wk)
* Use of prescription medications at the time of the study that directly affect endpoints of interest (e.g. hyperlipidemia, glycemic control, steroids, statins, anti-inflammatory agents, and over-the-counter weight loss aids)
* Current participation in another research study
* Less than 18 and over 39 years old
* BMI less than 18.5 and above 29.9 kg/m²
* Has HIV/AIDS or another disease that affects the immune system
* Unable to fast for 12 hours
* Gives regular blood donations and is unwilling to stop during the study
* Has monocytosis (>0.8 x 10³/microliter) or other abnormalities in hematologic parameters based on a screening complete blood count (CBC) with differential

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2023-11-14 (Actual); Primary Completion 2024-10-11 (Actual); Study Completion 2024-10-11 (Actual)

PRIMARY OUTCOMES:
Change in Monocyte subsets | Measured from samples taken at 0 hours (fasting) and 6 hours (postprandial) on 2 test days
  Monocyte subsets will be analyzed using flow cytometry. Subset analysis will be performed by labeling immune cells with anti-cluster of differentiation antigen 45 (anti-CD45), cluster of differentiation antigen 91 (anti-CD91), anti-CD14, and anti-CD16 fluorescently labeled antibodies.

SECONDARY OUTCOMES:
Change in white blood cell count | Measured from samples taken at 0 hours (fasting) and 6 hours (postprandial) on 2 test days
  White blood cell (WBC) count will be measured by a DxH 520 Hematology analyzer.
Change in lymphocyte count | Measured from samples taken at 0 hours (fasting) and 6 hours (postprandial) on 2 test days
  Lymphocyte (LY) count will be measured by a DxH 520 Hematology analyzer.
Change in monocyte count | Measured from samples taken at 0 hours (fasting) and 6 hours (postprandial) on 2 test days
  Monocyte (MO) count will be measured by a DxH 520 Hematology analyzer.
Change in change in neutrophil granulocyte count | Measured from samples taken at 0 hours (fasting) and 6 hours (postprandial) on 2 test days
  Neutrophil granulocyte (NE) count will be measured by a DxH 520 Hematology analyzer.
Change in eosinophil count | Measured from samples taken at 0 hours (fasting) and 6 hours (postprandial) on 2 test days
  Eosinophil (EO) count will be measured by a DxH 520 Hematology analyzer.
Change in basophil count | Measured from samples taken at 0 hours (fasting) and 6 hours (postprandial) on 2 test days
  Basophil (BA) count will be measured by a DxH 520 Hematology analyzer.
Change in red blood cell count | Measured from samples taken at 0 hours (fasting) and 6 hours (postprandial) on 2 test days
  Red blood cell (RBC) count will be measured by a DxH 520 Hematology analyzer.
Change in hemoglobin | Measured from samples taken at 0 hours (fasting) and 6 hours (postprandial) on 2 test days
  Hemoglobin (HGB) will be measured by a DxH 520 Hematology analyzer.
Change in hematocrit | Measured from samples taken at 0 hours (fasting) and 6 hours (postprandial) on 2 test days
  Hematocrit (HCT) will be measured by a DxH 520 Hematology analyzer.
Change in mean corpuscular volume | Measured from samples taken at 0 hours (fasting) and 6 hours (postprandial) on 2 test days
  Mean corpuscular volume (MCV) will be measured by a DxH 520 Hematology analyzer.
Change in mean corpuscular hemoglobin | Measured from samples taken at 0 hours (fasting) and 6 hours (postprandial) on 2 test days
  Mean corpuscular hemoglobin (MCH) will be measured by a DxH 520 Hematology analyzer.
Change in mean corpuscular hemoglobin concentration | Measured from samples taken at 0 hours (fasting) and 6 hours (postprandial) on 2 test days
  Mean corpuscular hemoglobin concentration (MCHC) will be measured by a DxH 520 Hematology analyzer.
Change in red blood cell distribution width | Measured from samples taken at 0 hours (fasting) and 6 hours (postprandial) on 2 test days
  Red blood cell distribution width (RDW) will be measured by a DxH 520 Hematology analyzer.
Change in red blood cell distribution width standard deviation | Measured from samples taken at 0 hours (fasting) and 6 hours (postprandial) on 2 test days
  Red blood cell distribution width standard deviation (RDW-SD) will be measured by a DxH 520 Hematology analyzer.
Change in platelet count | Measured from samples taken at 0 hours (fasting) and 6 hours (postprandial) on 2 test days
  Platelet (PLT) count will be measured by a DxH 520 Hematology analyzer.
Change in mean platelet volume | Measured from samples taken at 0 hours (fasting) and 6 hours (postprandial) on 2 test days
  Mean platelet volume (MPV) will be measured by a DxH 520 Hematology analyzer.
Change in CD45 gene expression | Measured from samples taken at 0 hours (fasting) and 6 hours (postprandial) on 2 test days
  Transcriptional changes in non-classical and classical monocytes will be measured by RNA-sequencing following the isolation of non-classical monocytes from peripheral blood by fluorescence-activated cell sorting (FACS) using anti-CD45 fluorescently labeled antibodies.
Change in CD91 gene expression | Measured from samples taken at 0 hours (fasting) and 6 hours (postprandial) on 2 test days
  Transcriptional changes in non-classical and classical monocytes will be measured by RNA-sequencing following the isolation of non-classical monocytes from peripheral blood by fluorescence-activated cell sorting (FACS) using anti-CD91 fluorescently labeled antibodies.
Change in CD14 gene expression | Measured from samples taken at 0 hours (fasting) and 6 hours (postprandial) on 2 test days
  Transcriptional changes in non-classical and classical monocytes will be measured by RNA-sequencing following the isolation of non-classical monocytes from peripheral blood by fluorescence-activated cell sorting (FACS) using anti-CD14 fluorescently labeled antibodies.
Change in CD16 gene expression | Measured from samples taken at 0 hours (fasting) and 6 hours (postprandial) on 2 test days
  Transcriptional changes in non-classical and classical monocytes will be measured by RNA-sequencing following the isolation of non-classical monocytes from peripheral blood by fluorescence-activated cell sorting (FACS) using anti-CD16 fluorescently labeled antibodies.
Change in expression of very late antigen-4 | Measured from samples taken at 0 hours (fasting) and 6 hours (postprandial) on 2 test days
  Monocyte adhesion molecule expression of very late antigen-4 (VLA-4) will be assessed using flow cytometry.
Change in expression of C-X3-C motif chemokine receptor 1 | Measured from samples taken at 0 hours (fasting) and 6 hours (postprandial) on 2 test days
  Monocyte adhesion molecule expression of C-X3-C motif chemokine receptor 1 (CX3CR1) will be assessed using flow cytometry.
Change in expression of Notch2 | Measured from samples taken at 0 hours (fasting) and 6 hours (postprandial) on 2 test days
  Monocyte adhesion molecule expression of Notch2 will be assessed using flow cytometry.
Change in expression of colony stimulating factor 1 receptor | Measured from samples taken at 0 hours (fasting) and 6 hours (postprandial) on 2 test days
  Monocyte adhesion molecule expression of colony stimulating factor 1 receptor (CSFR1) will be assessed using flow cytometry.
Change in expression of scavenger receptor class B, member 3 | Measured from samples taken at 0 hours (fasting) and 6 hours (postprandial) on 2 test days
  Monocyte adhesion molecule expression of scavenger receptor class B, member 3 (CD36) will be assessed using flow cytometry.
Change in intensity of filamentous-actin | Measured from samples taken at 0 hours (fasting) and 6 hours (postprandial) on 2 test days
  Filamentous-actin (F-actin) intensity will be assessed using phalloidin.
Change in levels of interleukin-6 | Measured from samples taken at 0 hours (fasting) and 6 hours (postprandial) on 2 test days
  Plasma markers of systemic inflammation including interleukin-6 will be measured by ELISA.
Change in levels of interleukin-8 | Measured from samples taken at 0 hours (fasting) and 6 hours (postprandial) on 2 test days
  Plasma markers of systemic inflammation including interleukin-8 will be measured by ELISA.
Change in levels of C-reactive protein | Measured from samples taken at 0 hours (fasting) and 6 hours (postprandial) on 2 test days
  Acute phase reactants including C-reactive protein (CRP) will be measured by ELISA.
Change in levels of serum amyloid A | Measured from samples taken at 0 hours (fasting) and 6 hours (postprandial) on 2 test days
  Acute phase reactants including serum amyloid A (SAA) will be measured by ELISA.
Change in levels of chemokine ligand 2 | Measured from samples taken at 0 hours (fasting) and 6 hours (postprandial) on 2 test days
  Chemokines including chemokine ligand 2 will be measured by ELISA.
Change in levels of 8-isoprostane F2alpha | Measured from samples taken at 0 hours (fasting) and 6 hours (postprandial) on 2 test days
  Plasma markers of oxidative stress including 8-isoprostane F2alpha will be measured by ELISA.
Change in soluble cluster of differentiation antigen 146 | Measured from samples taken at 0 hours (fasting) and 6 hours (postprandial) on 2 test days
  Endothelial activation including soluble cluster of differentiation antigen 146 (CD146) will be measured by ELISA.
Change in levels of triglycerides | Measured from samples taken at 0 hours (fasting) and 6 hours (postprandial) on 2 test days
  Lipid-related markers including triglycerides will be measured by auto-analyzer, Cobas Integra 400+ instrument
Change in levels of total cholesterol | Measured from samples taken at 0 hours (fasting) and 6 hours (postprandial) on 2 test days
  Lipid-related markers including total cholesterol will be measured by auto-analyzer, Cobas Integra 400+ instrument
Change in levels of HDL-cholesterol | Measured from samples taken at 0 hours (fasting) and 6 hours (postprandial) on 2 test days
  Lipid-related markers including HDL-cholesterol (HDL-C) will be measured by auto-analyzer, Cobas Integra 400+ instrument
Change in levels of LDL-cholesterol | Measured from samples taken at 0 hours (fasting) and 6 hours (postprandial) on 2 test days
  Lipid-related markers including LDL-cholesterol (LDL-C) will be measured by auto-analyzer, Cobas Integra 400+ instrument
Change in levels of glucose | Measured from samples taken at 0 hours (fasting) and 6 hours (postprandial) on 2 test days
  Plasma glucose will be measured by auto-analyzer, Cobas Integra 400+ instrument

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Snodgrass, PhD, Principal Investigator — USDA, Western Human Nutrition Research Center
Locations (1):
- USDA Western Human Nutrition Research Center, Davis, California, United States

IPD SHARING:
Plan to Share IPD: No